CLINICAL TRIAL: NCT03903731
Title: Safety and Performance of Journey II BCS Total Knee System. A Retrospective, Multicenter Study. Patient Reported Outcomes Measures
Brief Title: Safety and Performance of Journey II BCS Total Knee System Patient Reported Outcome Measures
Acronym: JIIPROMS
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-4049-08B
Record Dates: First submitted 2019-03-26; First posted 2019-04-04 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Journey II BCS Total Knee System
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Total knee arthroplasty with Journey II BCS Total Knee System — Journey II BCS Total Knee System

SUMMARY:
Safety and Performance of Journey II BCS Total Knee System. A Retrospective, Multicenter Study. Patient Reported Outcome Measures.

ELIGIBILITY:
Inclusion Criteria:

* Subject received primary uni- or bi-lateral total knee arthroplasty with the Journey II BCS Total Knee System for approved indication;
* The TKA occurred at least 12 weeks prior to enrollment
* Subject records contain Patient Reported Outcome data obtained ≤3 months prior to as well as ≥6 months post-enrollment.

Exclusion Criteria:

* Subject received the JOURNEY II BCS Total Knee System on the affected knee as a revision for a previously failed total or unicondylar knee arthroplasty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who received the Journey II BCS Total Knee System
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Revision of one or more study device components | Implantation through study completion, approximately 8 years
  We are measuring the number of revision cases

SECONDARY OUTCOMES:
Health care utilization: Rehabilitation | Implantation through study completion, approximately 8 years
  Number of sessions and duration of rehabilitation in weeks
Return to Work | Implantation through study completion, approximately 8 years
  Changes in employment status will be recorded with the date on which the change occurred and the change status.
Knee Society Score (KSS) | Baseline through last study visit, approximately 8 years
  Knee Society Score (KSS), a physician- and self-administered questionnaire consisting of several items to measure the outcomes; in this study, the following KOOS scores ranging from 0 to 100 were analyzed: Symptoms Score, Satisfaction Score, Expectation Score, Walking and Standing Score, Standard Activity Score, Advanced Activity Score, Discretionary Activity Score, and Functional Activities Score. Lower KSS scores indicated worse knee conditions.
Visual Analogue Scale (VAS) | Baseline through last study visit, approximately 8 years
  Visual Analogue Scale (VAS), a self-administered psychometric response instrument to evaluate subject-reported assessment of pain in each knee. There are multiple ways to present VAS scores; in this study, the numerical score ranged from 0 to 100 was used, with the higher score corresponding to the worse pain.
Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index | Baseline through last study visit, approximately 8 years
  The Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index, a self-administered questionnaire consisting of several items (grouped into symptoms, function, daily living, pain, etc) to measure the outcomes using the scores: Total WOMAC score (sum of all scores), WOMAC pain score (range 0 to 20), WOMAC stiffness score (range 0 to 8), and WOMAC physical function score (range of 0 to 68). The higher WOMAC scores corresponded to worse outcomes.
Total Knee Assessment Score | Baseline through last study visit, approximately 8 years
  Total Knee Assessment score is a self-administered questionnaire comprising multiple-choice questions regarding subjects' knee-related pain and limitations in ability to work, sports, and other daily living activities. In this study, the numbers and percentages of subjects answering each multiple-choice question were summarized. The higher percentage of subjects giving an answer indicating a higher level of limitations was indicative of worse outcomes.
Oxford Knee Assessment (OKS) | Baseline through last study visit, approximately 8 years
  Oxford Knee Assessment (OKS) is a self-administered questionnaire comprising multiple-choice questions aimed to grade subjects' ability to perform daily activities. The overall score is the sum of all items and range from 0 to 48, with a higher score corresponding to better outcomes.
Knee Injury and Osteoarthritic Outcome Score (KOOS) | Baseline through last study visit, approximately 8 years
  Knee Injury and Osteoarthritic Outcome Score (KOOS) is a self -administered joint-specific questionnaire comprising questions regarding subject's symptoms, knee stiffness, pain, function and daily living, function and sports and recreational activities, and quality of life; in this study, the following KOOS scores ranging from 0 to 100 (with a score of 0 indicating the worst possible symptoms) were analyzed: Pain Score, Other Symptoms Score, Function in Daily Living Score, Function in Sport and Recreation Score, and Quality of Life Score.
Knee Injury and Osteoarthritic Outcome Score Jr (KOOS Jr) | Baseline through last study visit, approximately 8 years
  Knee Injury and Osteoarthritic Outcome Score Jr (KOOS Jr) is a shorter self-administered alternative to KOOS focusing on joint pain, stiffness, and daily living and allowing for faster completion by the subject. In this study, the KOOS Interval Score ranging from 0 to 100 was analyzed (with a score of 0 indicating the worst possible symptoms).
SF-12 Version 1 | Baseline through last study visit, approximately 8 years
  SF-12 Version 1 is a self-administered multipurpose (not aimed to specific disease group) short form survey with questions selected from the longer SF-36 Health Survey and comprising the following scores: Physical Health Composite Score (range 0 for the worst health to 100 for the best health) and Mental Health Composite Score (range 0 for the worst health to 100 for the best health)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Dayton, MD, Principal Investigator — Department of Orthopaedics, University of Colorado Denver; David J. Mayman, MD, Principal Investigator — Hospital for Special Surgery, New York; Harold E. Cates, MD, Principal Investigator — Tennessee Orthopaedic Clinics; Hilde Vandenneucker, MD, Principal Investigator — UZ Leuven; Peter Black, MBBCh, Principal Investigator — Anglesea Clinic Orthopaedics
Locations (5):
- United States (3):
  - Department of Orthopaedics, University of Colorado Denver, Aurora, Colorado
  - Hospital for Special Surgery, New York, New York
  - Tennessee Orthopaedic Clinics, Knoxville, Tennessee
- UZ Leuven, Leuven, Belgium
- Anglesea Clinic Orthopaedics, Hamilton, New Zealand

IPD SHARING:
Plan to Share IPD: No